CLINICAL TRIAL: NCT07033884
Title: Reducing Firearm Suicide Among Veterans: Evaluating the Effectiveness of Peer-Delivered Lethal Means Counseling
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MHBC-003-24F; 1 IK2 CX002877-01A1 (Other Grant/Funding Number: VA Office of Research & Development)
Record Dates: First submitted 2025-06-09; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Suicide; Secure Firearm Storage
Keywords: Suicide Prevention; Firearms; Motivational Interviewing
MeSH Terms: conditions — Suicide; Suicide Prevention | interventions — Safety

STUDY DESIGN:
Intervention Model Description: Participants are randomized (1:1) upon enrollment to one of two conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PEERS (Experimental): Veterans in this condition will complete the PEERS intervention and will receive the same psychoeducational materials as the active control group.
  Interventions: Behavioral: Peer Engagement and Exploration of Responsibility and Safety
- Active Control (Other): Veterans in this condition will receive psychoeducational materials on lethal means safety and will have NO interaction with peers.
  Interventions: Other: Active Control

INTERVENTIONS:
Behavioral: Peer Engagement and Exploration of Responsibility and Safety — PEERS involves a one-on-one session with a firearm-owning Veteran peer interventionist. The appointment will last between 15 minutes and one hour, and the modality (i.e., in-person or virtual) will be based on Veteran participant preference. Principal components of the PEERS session will include: 1) engaging - initiating conversation in a non-confrontational manner; 2) focusing - quickly concentrating the discussion on the topic of firearms and means safety; 3) evoking - reflecting the participants' reasons both for and against engaging in means safety, leveraging the participants' own rationale for change as a tool for increasing behavior change; and 4) planning - once a plan is agreed upon, this information is put into writing. Participants will also be provided the same psychoeducational materials provided to the participants in the active control condition.
  Other Names: PEERS
  Arms: PEERS
Other: Active Control — Veterans will receive no treatment and will not interact with peers. A no treatment control condition was selected due to the preventative nature of PEERS, as well as the early stage of evaluation for this intervention. However, given the varied recruitment outlets and subsequent lack of standardized "usual care," as well as ethical concerns with not providing important resources to firearm owning Veterans, two informational handouts will be added to this control condition. Specifically, Veterans in this condition will be provided with an informational handout developed by the National Sports Shooting Foundation, which includes a variety of secure firearm storage options, as well as a handout listing national mental health and suicide prevention resources.
  Other Names: AC
  Arms: Active Control

SUMMARY:
Suicide prevention is a top priority for the Department of Veterans Affairs (VA), with a major emphasis on developing innovative and effective ways to prevent firearm suicide. Research suggests that secure firearm storage can decrease risk for suicide and the current project aims to evaluate a novel approach to increasing secure storage through an experimental design. The intervention takes one-hour or less and involves a peer-to-peer discussion about secure firearm storage, focusing on participants' reasons for and against using more secure firearm storage practices. The project will evaluate whether Veterans who receive this intervention report greater use of secure firearm storage practices than Veterans who receive only psychoeducational materials on this topic. Secure firearm storage practices will be evaluated over the course of one year. It is hypothesized that Veterans who engage in the peer-to-peer intervention will report greater use of secure firearm storage practices than those who receive only psychoeducational materials. Relevant to Veterans' health, secure firearm storage decreases Veteran firearm suicide risk and may help prevent suicide. In addition, this peer-delivered intervention is preferred by Veterans, and has the flexibility to be implemented before suicide risk develops and in settings outside of the VA. This means the intervention has the potential to reach more Veterans, even those who do not receive VA healthcare.

DETAILED DESCRIPTION:
Veterans die by suicide at a rate 1.72 times greater than civilian counterparts. Notably, 72% of Veteran suicides result from a firearm, making firearm suicide prevention a leading priority for the Department of Veterans Affairs (VA). Secure firearm storage (e.g., unloaded, locked) mitigates risk of firearm suicide, but these practices are uncommon among firearm owning Veterans. Lethal means counseling (LMC), an intervention that promotes reduced access to potentially lethal suicide methods (e.g., firearms) through one-on-one interactions, is a promising approach to promoting secure firearm storage among Veterans. However, there are limitations to the reach and acceptability of LMC among firearm owning Veterans within VA, including healthcare providers' limited time during appointments and firearm owners' stated preference to discuss firearms with those perceived to be credible, such as fellow Veterans. As a result, most Veteran firearm owners, including those with recent suicidal ideation, report that they have not discussed firearm access with their healthcare providers. It is crucial to expand LMC efforts to non-clinician messengers to reach more Veterans. What remains unknown is how effective preferred messengers are in changing firearm storage behaviors, as well as what mechanisms impact or account for subsequent changes in firearm storage behaviors. Thus, there is a critical need to evaluate the effectiveness of peer-delivered LMC among Veteran firearm owners. Without such knowledge, preventing suicide within this population will likely remain difficult.

The overall objective of the current study is to estimate the effectiveness, as well as factors that impact or account for the effectiveness, of peer-delivered LMC. My central hypothesis is that peer-delivered LMC will lead to greater use of secure firearm storage and this will be accounted for and influenced by mechanisms conceptualized by the Theory of Planned Behavior (TPB), those proposed to be relevant in prior research, and unique mechanisms that have yet to be identified. This hypothesis was formulated on the basis of preliminary data generated through a Clinical Sciences Research and Development Career Development Award-1. During that study, I adapted a healthcare provider-delivered LMC intervention, found to increase secure firearm storage among National Guard members, for peer-delivery through an expert panel. The resulting intervention, Peer Engagement and Exploration of Responsibility and Safety (PEERS), is a 15-60 minute one-on-one LMC session centered around Motivational Interviewing principles and delivered by Veterans. In a single arm pilot trial, PEERS was feasible and acceptable among Veteran firearm owners. Thus, the rationale for this project is to determine the effectiveness, as well as mechanisms that impact or account for the effectiveness, of PEERS, providing new opportunities for suicide prevention among Veteran firearm owners. Two specific aims are proposed:

1. Estimate the superiority of PEERS compared to a psychoeducation control condition on secure firearm storage in a randomized controlled trial (N = 100; 1:1). My working hypothesis is Veterans receiving PEERS will demonstrate greater use of secure firearm storage than Veterans in the psychoeducation condition.
2. Identify indirect (2a & 2c) and moderating (2b & 2c) effects of the relationship between PEERS and secure firearm storage. My working hypothesis, based on the TPB, is that changes in secure firearm storage will be indirect through attitudes towards secure firearm storage, subjective norms about secure firearm storage, perceived ease of changing firearm storage, and intentions to change firearm storage (2a). I further hypothesize, based on prior research, that primary motivation for ownership (personal/family protection), Posttraumatic Stress Disorder hyperarousal symptoms, and low belief in the relationship between firearms and suicide risk, will attenuate changes in secure firearm storage (2b). To identify other factors that may influence the relationship between PEERS and secure firearm storage, I will recruit up to 24 Veterans who participated in PEERS for individual qualitative interviews regarding barriers and facilitators to engagement in the intervention (2c).

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* Owns at least one personal firearm
* Displays some level of unsecure firearm storage (i.e., scores < 6 on MIRECC Lethal Means Questionnaire eligibility screener)
* Capable of meeting via virtual modalities for appointments (i.e., owns a device capable of connecting for virtual appointments, has internet access)

Exclusion Criteria:

* Active psychosis
* Insufficient English language skills
* No reliable access to a telephone and/or device for attending appointments via virtual modalities
* Prior participation in the PI's CDA-1 study (N = 16)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2029-05-31 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Modified MIRECC Lethal Means Questionnaire | Eligibility Screening, Baseline, Follow-ups (1-week, 6-months, 1-year)
  The MIRECC Lethal Means Questionnaire (Simonetti, 2017) is a 13-item self-report measure designed to assess experiences with firearms. Items include questions about number and type of firearms owned, primary reason for firearm ownership, and firearm handling. It also includes items related to firearm storage practices. Two open-ended questions were also added to allow participants to describe, in their own words, their current firearm storage practices, and at follow-ups to describe any changes they've made to their firearm storage that is not captured in the other questions. Responses to three key firearm storage items will be totaled to create a composite storage score, with higher scores indicating safer storage practices. Range of values: 0-6.
Theory of Planned Behavior | Baseline and Follow-ups (1-week, 6-months, 1-year)
  A 15-item measure was designed using Francis and colleagues' (2004) guide to assess each of the four subdomains of the Theory of Planned Behavior. Specifically, there are three items assessing intentions to increase secure firearm storage (e.g., "I intend to increase my use of secure firearm storage"), four items assessing attitudes towards increasing secure firearm storage, four items assessing subjective norms surrounding increasing secure firearm storage (e.g., "People who are important to me want me to increase my use of secure firearm storage"), and four items assessing perceived behavioral control of increasing secure firearm storage. All items include 7-point Likert scale response options and the items within subdomains (e.g., intentions, attitudes) are averaged to produce overall subdomain scores. Range of values: 1-7.
Beliefs and Attitudes about Firearms and Suicide | Baseline and Follow-ups (1-week, 6-months, 1-year)
  A 3-item questionnaire used to evaluate belief in relationships related to suicide risk. Items include, "To what extent do you think owning a firearm is related to suicide risk?", "To what extent do you think how a firearm is stored (e.g., gun safe, loaded) is related to suicide risk?", and "To what extent do you agree with the statement 'if somebody wants to die by suicide and you prevent them from using a specific method, they will simply find another way to die'?" Participants will respond on a 5-point Likert scale, with higher scores indicating higher belief in the statement or described relationship. Range of values: 0-12.
Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | Baseline and Follow-ups (1-week, 6-months, 1-year)
  PTSD symptoms will be assessed using the PCL-5, including the criterion A face page (Blevins et al., 2015). The PCL-5 includes a brief set of questions assessing whether an individual has experienced a criterion A stressor, followed by a 20-item self-report questionnaire designed to assess each of the 20 Diagnostic and Statistical Manual of Mental Disorders - 5th Edition (DSM-5) PTSD symptoms. Participants will first be asked to respond to five questions on the face page assessing for criterion A stressors. Next, they will be asked to respond to the 20-item self-report measure using a 5-point Likert scale, with higher scores suggesting higher symptom severity. In addition to a total score, the PCL-5 yields four subscale scores reflecting the four PTSD symptom clusters (i.e., re-experiencing, avoidance, alteration in cognitions and mood, and arousal and reactivity). Range of values: 0-80.

SECONDARY OUTCOMES:
Semi-Structured Interview | Post 1-year Follow-up
  Qualitative feedback on barriers and facilitators to engagement in PEERS will be obtained through audio-recorded semi-structured interviews with up to 24 Veterans who were randomized to the PEERS condition. In addition to self-generated barriers and facilitators to engagement in PEERS, Veterans will be asked to identify non-VHA settings in which they may prefer to receive such an intervention. The semi-structured interview template was adapted from Dobscha et al., 2021.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Houtsma, PhD, Principal Investigator — Southeast Louisiana Veterans Health Care System, New Orleans, LA
Locations (1):
- Southeast Louisiana Veterans Health Care System, New Orleans, LA, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No